CLINICAL TRIAL: NCT02789748
Title: PErsonalized and Adaptive Kinesthetic stImulation Therapy, Based on Cardio-respiratory Holter moNitoring, for Sleep Apnea syndrOmes
Acronym: EKINOx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LivaNova (Industry)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IAHO03
Record Dates: First submitted 2016-02-18; First posted 2016-06-03 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment ON (Experimental): Kinesthetic stimulation administered during one night
  Interventions: Device: Kinesthetic stimulation
- Treatment OFF (No Intervention): NO kinesthetic stimulation administered during one night

INTERVENTIONS:
Device: Kinesthetic stimulation — Activation of mechanoreceptors by vibration bursts
  Arms: Treatment ON

SUMMARY:
This study aims at quantifying the performance of kinesthetic stimulation to reduce the burden of obstructive sleep apneas and hypopneas.

DETAILED DESCRIPTION:
Severe sleep apnea patients will undergo two polysomnographies (PSG), one with kinesthetic stimulation triggered on the detection of apneas and hypopneas (treated night ) and the other without kinesthetic stimulation (non-treated night ). Comparison of apnea and hypopnea indices (AHI) and of oxygen saturation between the treated and non-treated night will be taken as indicators to quantify the performance of this potential new therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following criteria at the time of enrollment may be included:

* Man or woman aged more than 18 years old.
* Patient with severe obstructive apnea syndrome diagnosed on polysomnography or polygraphy performed less than 6 months ago with (AHI > 30/h and 80% of obstructive events) and (ODI 4% > 20 or time with SaO2 below 90% > 5%).
* Patient free from continuous positive airway pressure (CPAP) treatment or any other SAS treatment for at least 3 months
* Patient with no psychrotropic medication or stable psychotropic medication since the diagnostic polysomnography or polygraphy examination
* Patient was informed and has signed the informed consent

Exclusion Criteria:

Patients who meet any one of these criteria will be excluded from the study:

* Patients sleeping less than 4 hours per night
* Patients suffering from respiratory failure, such as chronic obstructive pulmonary disease (COPD), pneumonia, pulmonary edema, pulmonary fibrosis, asthma, pulmonary arterial hypertension.
* Patients developing periodic breathing or Cheyne Stokes respiration
* Obese patient (BMI>35kg/m2)
* Patient with autonomic dysfunction (symptoms include orthostatic hypotension, exercise intolerance, sweating abnormalities, digestion difficulties, urinary problems, vision problems) as complication of diabetes, Parkinson's disease or other primary pathologies.
* Patient suffering from restless leg syndrome or periodic leg movement (PLM) not related to obstructive sleep apnea, i.e. PLM index > 15/h excluding movements linked to respiratory events.
* Patient suffering from positional sleep apnea syndrome (SAS), i.e. supine apnea hypopnea index (AHI) at least twice that of the non-supine AHI
* Patient suffering from severe peripheral neuropathy
* Vulnerable patient in accordance with article L1121-6 of Code de la Santé Publique (CSP)
* Patient already involved in another clinical study that could affect the result of this study
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Rate of responder to the therapy | Day 1 post-discharge
  A patient is defined as 'responder' to the therapy by comparison of the treated night to the non-treated night based on:
  * The oxygen desaturation index (ODI)
  * The time spent below 90% of oxygen saturation or
  * The apnea hypopnea index (AHI) reduction

SECONDARY OUTCOMES:
Adverse device effect | Day 1 post-discharge
  Adverse Events related to the investigational device
Effect on apneas/hypopneas duration | Day 1 post-discharge
  Therapy effect on shortening respiratory events
Effect on modified apnea hypopnea index | Day 1 post-discharge
  The modified apnea hypopnea indices (AHIs) will be compared between the treated and non-treated night and defined based on the duration of the respiratory disorders
Instantaneous heart rate measurement (bpm) during the night ON and the night OFF | Day 1 post-discharge
Number of arousals per night - comparison night ON and night OFF | Day 1 post-discharge
  The micro-arousal index will be calculated on the polysomnography recording.
Effect on an objective measure of somnolence (Osler) | Day 1 post-discharge
  Osler test (optional) performed after treated night and non-treated night

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hospital Beziers, Béziers
  - University Hospital Grenoble, Grenoble
  - CHU Rennes, Rennes
  - University Hospital Tours, Tours